CLINICAL TRIAL: NCT05915169
Title: Investigation of the Effects of Topical Haemoglobin Wound Care Spray in Pressure Ulcer Care
Brief Title: The Effects of Topical Haemoglobin Spray in Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: Abant Izzet Baysal University (Other); Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Özge Uçar, Research Assistant, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-OU-01
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pressure Ulcer; Wound Heal
Keywords: pressure ulcer; nursing care; topical haemoglobin spray; wound dressing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: topical haemoglobin spray care group and standart gas dressing with saline solution care group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical haemoglobin spray care group (Experimental): Patients with stage 2 pressure ulcers in the sacrum area will be treated with topical haemoglobin spray every 3 days for 2 months.
  Interventions: Other: Topical haemoglobin wound care spray
- group of gas dressings with saline solution (No Intervention): Patients with stage 2 pressure ulcers in the sacrum area will receive routine saline gas dressing for 2 months.

INTERVENTIONS:
Other: Topical haemoglobin wound care spray — It is a wound care spray used in the care of chronic wounds.
  Arms: topical haemoglobin spray care group

SUMMARY:
A prospective randomised controlled experimental study was planned to compare the effects of pressure sore dressing using topical haemoglobin and traditional gauze dressing using saline on the healing process and cost of pressure sores in patients with pressure sores.

DETAILED DESCRIPTION:
Pressure sores are a serious health problem because they increase mortality, decrease quality of life, prolong hospital stays, increase patient care costs, impair body image, prolong the healing process, and have many other negative effects.

The European Pressure Ulcer Advisory Panel (EPUAP), National Pressure Ulcer Advisory Panel (NPIAP), and Pan Pacific Pressure Ulcer Association (PPPIA) 2019 guidelines report that the prevalence of pressure ulcers in healthcare settings ranges from 10% to 72.5%, with large variations between different clinics and geographies. In the United States, the cost of pressure sore treatment to organisations is estimated to be $11 billion annually. Pressure sores will continue to be an important public health problem today and in the future, especially due to the increasing number of elderly people in the world and in our country, chronic diseases, comorbidity, and palliative conditions.

Therefore, the study was planned as a prospective randomised controlled experimental trial to compare the effects of pressure sore dressing using topical haemoglobin and traditional gauze dressing using saline on the healing process and cost of pressure sores in patients with pressure sores.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years of age,
2. Normal albumin and protein levels,
3. Stage 2 pressure ulcer,
4. Blood glucose level is within normal limits,
5. the consent of the patient himself or his guardian.

Exclusion Criteria:

1. being under 18 years of age,
2. Pressure ulcers in areas other than the sacrum,
3. Stage 1, Stage 3, Stage 4, unstageable pressure ulcers,
4. Albumin and protein values are lower than normal,
5. Blood glucose level is not within normal limits,
6. the patient himself/herself or his/her guardian does not authorise it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer scale for healing | 2 months
  PUSH is an acronym for Pressure Ulcer Scale for Healing. The National Pressure Ulcer Advisory Panel developed this tool to monitor pressure healing over time. The PUSH Tool monitors three parameters: surface area of the wound, wound exudate, and type of wound tissue. Wounds are measured using a centimeter ruler. The scores are rated from 0 to 10 according to the size of the wound.

SECONDARY OUTCOMES:
cost chart | 2 months
  The researcher has been formed by the researchers. The materials used for 2 months will be recorded in this table with their quantity. At the end of the study, cost calculation will be made based on current prices.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Uçar, Phd scholar, Principal Investigator — Research Assisstant
Locations (1):
- Bartın Üniversitesi, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No